CLINICAL TRIAL: NCT03384862
Title: Nutrition, Arsenic and Cognitive Function in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Mary Gamble, Associate Professor of Environmental Health Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AAAQ9290; 2P42ES010349-16 (NIH)
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Arsenic Exposure
Keywords: Arsenic exposure
MeSH Terms: interventions — Vitamin B 12; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participants, field staff, and investigators will be blinded to the intervention status of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Intervention Arm (Experimental): 5 μg vitamin B12 plus 400 μg folic acid
  Interventions: Dietary Supplement: Vitamin B12; Dietary Supplement: Folic Acid
- Control Arm (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — 5 μg/d vitamin B12 to be given orally. This is a standard nutritional supplement commonly used in the US.
  Arms: Nutritional Intervention Arm
Dietary Supplement: Placebo — Placebo pills, with same appearance as intervention pills.
  Arms: Control Arm
Dietary Supplement: Folic Acid — 400 μg/d folic acid to be given orally. This is a standard nutritional supplement commonly used in the US.
  Arms: Nutritional Intervention Arm

SUMMARY:
The main goals of this study are to evaluate whether supplementation with folate and vitamin B12 to 8 to 10 year old children, in conjunction with reduction in arsenic exposure, can increase arsenic methylation and lower blood arsenic and blood monomethyl arsenic (as previously observed in adults). The investigators will also explore whether folate and B12 can mitigate arsenic-related decrements in cognitive abilities.

DETAILED DESCRIPTION:
While reducing arsenic (As) exposure in Bangladesh and the U.S. must continue to be a top priority, this has proven difficult. After decades of efforts to reduce exposure, 42 million people in Bangladesh remain exposed to As above 10 µg/L, the WHO guideline for As in drinking water. Risk for arsenic-related health outcomes lingers for decades after exposure has been reduced. Innovative strategies to lower arsenic exposure and and reduce its potential adverse health effects of As are needed.

ELIGIBILITY:
Inclusion Criteria:

* Age-eligible children of parents enrolled in the Health Effects of Arsenic Longitudinal Study cohort

Exclusion Criteria:

* siblings
* twins
* children who are not attending school
* children with known physical disability or known chronic illness

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 239 (Actual)
Dates: Start 2018-01-27 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Change in arsenic methylation | Up to 12 Weeks
  Change in arsenic methylation patterns in blood and urine. The ability to methylate arsenic influences an individual's ability to excrete it in urine.
Change in in blood arsenic | Up to 12 Weeks
  Change in arsenic level in blood is to be measured in mg/L. This is an indicator of the body burden of arsenic and arsenic excretion
Change in blood monomethyl arsenic | Up to 12 Weeks
  Change in monomethyl arsenic level in blood is to be measured in units of ug/L. This is an indicator of the body burden of arsenic and arsenic methylation capacity.

OTHER OUTCOMES:
Change in WASI-II cognitive function test score | Up to 12 Weeks
  An improvement in scores on a test of cognitive function after receiving dietary supplements represent potential partial mitigation of arsenic- and nutrition-related cognitive decrements. Wechsler Abbreviated Scale of Intelligence (WASI-II) is a screen of verbal, non-verbal, and general cognitive ability. Higher score indicates higher cognitive function. Scores on the WASI-II can range from below 70 (demonstrating cognitive deficiency) to above 200 (demonstrating incredible genius) - typical "normal" or "average" scores are between 90-100. Higher values indicate a better score in terms of cognitive outcome while lower values indicate a poorer score. An improvement on WASI-II test scores for these participants would be demonstrated in a higher score on this test after receiving the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mary V Gamble, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bae S, Kamynina E, Guetterman HM, Farinola AF, Caudill MA, Berry RJ, Cassano PA, Stover PJ. Provision of folic acid for reducing arsenic toxicity in arsenic-exposed children and adults. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD012649. doi: 10.1002/14651858.CD012649.pub2. PMID 34661903